CLINICAL TRIAL: NCT05323994
Title: Description of the Effectiveness and Tolerability of аgomelatine in the Treatment of Patients With Depression Occurred After SARS-CoV-2 Infection in the Daily Clinical Practice in Russia (TELESPHOR)
Brief Title: Effectiveness and Tolerability of аgomelatine in the Treatment of Patients With Depression After SARS-CoV-2 (TELESPHOR)
Acronym: TELESPHOR
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-20098-069-RUS
Record Dates: First submitted 2022-04-08; First posted 2022-04-12 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Depression; COVID-19
MeSH Terms: conditions — Depression; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-centre, observational, non-interventional study, which will prospectively collect clinical and socio-demographic data from patients with depression occurred after COVID 19 in real clinical settings during 8 weeks of treatment.

10 clinics and 10 of psychiatrists and neurologists across the country will participate in the study and it is estimated that each investigating physician will enroll 10 patients.

DETAILED DESCRIPTION:
A patient with depression occurred within 3 month period after onset of confirmed COVID 19 infection who has already been recommended to initiate antidepressive treatment with agomelatine will be asked to provide a consent to participate in the study and in case of consent is positive the patient will be invited for 3 more visits starting from the date of the inclusion in the study according to clinical practice. Therefore clinical parameters needed for describing effectiveness and tolerability of agomelatine treatment will be prospectively collected at each of these visits. Antidepressive treatment of enrolled outpatients can be modified by investigating psychiatrist or neurologist at any time of the observation if required.

Following visits are planned:

1. Inclusion Visit 0 (V0) - inclusion in the study
2. Follow up Visits 1-2 (V1-V2) - visits at week 2 and week 4 after V0.
3. Final Visit 3 (V3) - visit at week 8 after V0.

ELIGIBILITY:
Inclusion Criteria:

* Obtained signed informed consent from the patient.
* Age of 18-65 years old.
* Out-patient with confirmed COVID 19 infection within 3 months period before the date of inclusion.
* Confirmed depression with total HAMD-17 score of 8-24 required treatment with antidepressive medicines.
* Decision to administer agomelatine preceeds the decision to include a patient in the study.

Exclusion Criteria:

* Current participation in any clinical trial or during 30 day period from inclusion visit.
* Suicide risk (accoding clinical evaluation of investigator).
* Psychotics symptoms (according clinical evaluation of investigator).
* Schizophrenia, schizo-affective disorders, organic damages of CNS, dementia, epilepsy, multiple sclerosis, Parkinson disease, Alzeimert disease, Bipolar disorders.
* Alcohol abuse or drug addiction in anamnesis.
* Severe or decompensated somatic or neurological disorders.
* MAO inhibitors during last 2 weeks.
* Treatment by others psychotropic products (antipsychotics, anxiolitics etc.).
* Any contraindications to agomelatine in accordance to the local SmPC.
* Patients with severe/decompensated psychiatric, somatic or neurological disorders.
* Patients with any sign of liver failure (increase of transaminase up to 3 times higher), which needs to stop treatment with agomelatine.
* Patients who participate in any clinical trial or survey.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with depression occurred after COVID 19
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Autonomous Educational Institution of Higher Education "Peoples' Friendship University of Russia", Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Depression Occurred After COVID 19: Patients with the major depressive disorder (total score 8-24 on HAMD-17 - The Hamilton Rating Scale for Depression (HRSD), also called the Hamilton Depression Rating Scale (HDRS), sometimes also abbreviated as HAM-D, is a multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. It consists of 20 questions. For assessment of the severity of condition using a summary of total score where 0 - 7 "normal", 8 - 15 "mild depression",16 - 24 "moderate depression", 25 and more "severe depression" Depression treatment by agomelatine according to SMPC (Summary of Product Characteristics)
Period: Overall Study
Arm/Group | Patients With Depression Occurred After COVID 19
Started | 104
Completed | 103
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Depression Occurred After COVID 19
Number analyzed (Participants) | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 103
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 103

OUTCOME MEASURES:

1. Primary Outcome: Antidepressive Effectiveness of Agomelatine in Patients With Depression Episode Occurred After COVID-19 Assessed by HAMD-17 After 8 Weeks of Treatment in the Daily Clinical Practice.
Description: Mean change from baseline (BL) in total HAMD-17 (Hamilton Depression Rating Scale) score assessed at week 8 of the observational period.
  Assessment of the severity of condition using HAMD-17 (total score is reported, the total range from 0 to 51, where 0 score is no symptoms - 51 is for severe depression):
  0 - 7 "normal" (no marked symptoms of anxiety and depression), 8 - 15 "mild depression", 16 - 24 "moderate depression", 25 - 51 "severe depression"
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Depression Occurred After COVID 19
Number analyzed (Participants) | 103
score on a scale | 10.9 (4.90)

2. Secondary Outcome: Effectiveness of Agomelatine on Anxiety Symptoms Assotiated With the Depression and Assessed by HAMD-17 (Item 10 and Item 11) Baseline and 8 Weeks of Treatment of Patients Included in the Study.
Description: Mean change from baseline (BL) in HAMD-17 (Hamilton Depression Rating Scale) in item 10 (Psychic anxiety ) and item 11 (Somatic anxiety ) after 8 weeks of treatment of patients included in the study..
  Assessment of the severity in item 10:
  0- No difficulty
  1. Subjective tension and irritability
  2. Worrying about minor matters
  3. Apprehensive attitude apparent in face or speech
  4. Fears expressed without questioning
  Assessment of the severity in item 11:
  0- Absent
  1. Mild
  2. Moderate
  3. Severe
  4. Incapacitating
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Depression Occurred After COVID 19
Number analyzed (Participants) | 103
score on a scale
  item 10 | 0.5 (0.61)
  item 11 | 0.6 (0.56)

3. Secondary Outcome: Effectiveness of Agomelatine on Global Improvement and Social Functioning Assessed by CGI-I (Clinical Global Impression -Improvement) Score After 8 Weeks of Treatment of Patients Included in the Study.
Description: The clinical global impression - improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. The best is - "Very much improved" - 0 scores and "Very much worse"- 6 scores - is the worest
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Depression Occurred After COVID 19
Number analyzed (Participants) | 103
score on a scale | 1.3 (0.64)

4. Secondary Outcome: Effectiveness of Agomelatine on Quality of Life in Patients With Depression Episode Occurred After COVID-19 Assessed by SF-36 Questionnaire After 8 Weeks of Treatment of Patients Included in the Study.
Description: The Short Form (36) Health Survey (SF36 ) scale questioner was used. SF36 is is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Depression Occurred After COVID 19
Number analyzed (Participants) | 103
score on a scale
  physical component | 50.5 (5.70)
  mental component | 58.7 (6.91)

5. Secondary Outcome: Tolerability of Agomelatine After 8 Weeks of Treatment Based on Rate of Adverse Events Leading to Drug Discontinuation in Patients Included in the Study.
Description: Number of adverse events/ adverse drug reactions leading to drug discontinuation during the observational period.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Depression Occurred After COVID 19
Number analyzed (Participants) | 103
Participants | 1

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Patients With Depression Occurred After COVID 19
All-Cause Mortality (participants affected / at risk) | 0/103
Serious Adverse Events (participants affected / at risk) | 0/103
Other Adverse Events (participants affected / at risk) | 1/103
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Depression Occurred After COVID 19 (N=103)
inefficiency of treatment (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT05323994/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT05323994/ICF_001.pdf